CLINICAL TRIAL: NCT05723939
Title: Effects of Carnosine Supplementation in Form of Capsules and Functional Food on Cardiovascular Function
Brief Title: Carnosine Supplementation and Cardiovascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Principal investigator, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ZCICarnosine
Record Dates: First submitted 2023-01-22; First posted 2023-02-13 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Carnosine
Keywords: carnosine; oxidative stress; vascular reactivity; endothelium; inflammation; microcirculation; macrocirculation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carnosine (Experimental): Intake of carnosine supplement in form of capsules or functionally enriched chicken meet for three weeks
  Interventions: Dietary Supplement: Carnosine supplementation
- Control (Placebo Comparator): Intake of placebo capsules or regular chicken meet for three weeks
  Interventions: Dietary Supplement: Controls

INTERVENTIONS:
Dietary Supplement: Carnosine supplementation — Intake of carnosine supplement in form of capsules or functionally enriched chicken meet for three weeks
  Arms: Carnosine
Dietary Supplement: Controls — Intake of placebo capsules or regular chicken meet for three weeks
  Arms: Control

SUMMARY:
Carnosine is a dipeptide synthesized in the body from β-alanine and L-histidine. It was originally discovered in skeletal muscle where it is present in larger amounts than in other tissues, but it is also found in high concentrations in the brain, heart, and gastrointestinal tissues of humans. Although its physiological role has not been completely understood yet, carnosine is a non-enzymatic free-radical scavenger and a natural antioxidant and has anti-inflammatory and neuroprotective properties.

The hypothesis of this research is that the consumption of carnosine supplements in the form of capsules, as well as chicken meat enriched with carnosine (functional food) has a beneficial effect on vascular reactivity measured in different vascular basins, and the lipid profile with a positive effect on the reduction of oxidative stress and inflammatory response in healthy sedentary people. subjects and active athletes measured in different vascular basins.

The main goal of this study is to investigate the influence of carnosine supplement consumption (in the form of capsules and functional food) on vascular and endothelial function in a population of healthy young subjects and active athletes.

ELIGIBILITY:
Inclusion Criteria:

* young healthy sedentary individuals - did not perform regular physical activities for at least 12 months before conducting the study
* young healthy active athletes - have a minimum of 5 training sessions per week (mainly endurance training) for at least 12 months prior to conducting the study

Exclusion Criteria:

* smoking
* hypertension
* coronary disease
* diabetes
* hyperlipidemia
* kidney damage
* cerebrovascular and peripheral artery diseases
* and any other disease that could have an impact on vascular and endothelial function

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular endothelial function | 3 weeks
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to vascular occlusion (post occlusive reactive hyperaemia - PORH), in response to iontophoresis of acetylcholine (ACh) and local thermal hyperemia (LTH).
Macrovascular endothelial function | 3 weeks
  Measurement of flow mediated dilation (FMD) of brachial artery using ultrasound.
Cerebrovascular reactivity | 3 weeks
  Measurement of cerebrovascular blood flow using transcranial color Doppler (TCD).

SECONDARY OUTCOMES:
Lipid profile | 3 weeks
  Measurement of plasma cholesterol, HDL cholesterol, LDL cholesterol and triglycerides level.
Oxidative stress status | 3 weeks
  Measurement of Thiobarbituric Acid Reactive Substances (TBARS).
Systemic hemodynamics | 3 weeks
  Non-invasive assessment of systemic hemodynamics using impedance cardiography (CardioScreen 2000) - SV Stroke Volume (mL).
Serum Pro- and Anti-Inflammatory Cytokines, Chemokines, Growth Factors and Soluble Cell Adhesion Molecules Protein Concentration | 3 weeks
  Measurement of serum protein concentration (pg/mL) of various pro- and anti-inflammatory cytokines, chemokines, growth factors and soluble cell adhesion molecules by kits and panels for multiplex protein quantitation using the Luminex 200 instrument platform.
Body composition | 3 weeks
  Body composition and body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Fat Free Mass (FFM kg) and Fat (Fat Mass kg).
Body fluid status | 3 weeks
  Body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Total Body Water (TBW L), Extracellular Water (ECW L), Intracellular Water (ICW L), Plasma Fluid (PF L) and Interstitial Fluid (IF L).
Oxidative stress status | 3 weeks
  Measurement of Ferric-Reducing Ability of Plasma (FRAP).
Oxidative stress status | 3 weeks
  Measurement of enzyme activity assay of glutathione peroxidase (GPx).
Systemic hemodynamics | 3 weeks
  Non-invasive assessment of systemic hemodynamics using impedance cardiography (CardioScreen 2000) - CO Cardiac Output (L/min).
Systemic hemodynamics | 3 weeks
  Non-invasive assessment of systemic hemodynamics using impedance cardiography (CardioScreen 2000) - SVRI Systemic Vascular Resistance Index (dyn.s.cm-5 m2).

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Center of Excellence for Personalized Health Care, Josip Juraj Strossayer University of Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peric L, Drenjancevic I, Jukic I, Boris A, Susnjara P, Kolobaric N, Mihaljevic Z, Kralik Z, Kralik G, Kosevic M, Galovic O, Stupin A. Carnosine-enriched functional food enhances micro- and macrovascular endothelium-independent vasodilation in competitive athletes-a randomized study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-11. doi: 10.1139/apnm-2024-0458. PMID 39983097